CLINICAL TRIAL: NCT04151836
Title: Effect of Exercise Intervention on Body Composition and Quality of Life in Post-bariatric Surgery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 201901602A3
Record Dates: First submitted 2019-11-03; First posted 2019-11-05 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2020-10

CONDITIONS: Exercise
Keywords: Bariatric surgery; Body composition; Morbid obesity; Quality of life; Walking exercise
MeSH Terms: conditions — Motor Activity; Obesity, Morbid

STUDY DESIGN:
Intervention Model Description: Both groups were tested by demographic characteristics, dietary behavior measurement, SF-36 Questionnaire and body composition analyzer for the same project. The experimental group needs to cooperate with the moderate-intensity walking exercise training prescription for 3 times a week ; Control group no exercise intervention.
Who Masked: Outcomes Assessor
Masking Description: A statistician who did not participate in the study randomly assigned patients to the experimental or control group according to the list generated by the computer software.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- exercise group (Experimental): exercise education: A 12-week regimen of home-based walking exercises, include moderate intensity 30 minutes of exercise in week 1-4,40 minutes of exercise in 5-8 weeks,50 minutes in the 9-12 week,three times weekly in three month.We explained the participants how to perform the exercises, according to an instruction manual for the exercise regimen. Participants were instructed that the exercises would be effective only if they reached 65%-70% of the target Maximal heart rate(HRmax).
  Interventions: Other: Exercise education
- control group (No Intervention): These participants follows the standard post surgery follow-up consisting of counseling by dietitians, nurses and doctors.

INTERVENTIONS:
Other: Exercise education — weekly telephone or mobile application "LINE" consultations concerning exercise. we discussed whether participants' exercise fulfilled the prescribed intensity, duration, or frequency and whether the participants experienced any adverse effects.
  Arms: exercise group

SUMMARY:
This study will investigate the effectiveness of a rehabilitation program in improving body composition, and quality of life in patients with bariatric surgery in Taiwan.

Hypothesis:

1. The body composition in exercise group is significant improving than control group at 1 weeks, 1st, 2nd, and 3rd month.
2. The quality of life in exercise group is significant improving than control group at 1 weeks, 1st, 2nd, and 3rd month.

DETAILED DESCRIPTION:
This study will investigate the effectiveness of a rehabilitation program in improving body composition, and quality of life in patients with bariatric surgery in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

1. After the research purpose is stated, the subject agrees and is willing to participate in the researcher and is willing to sign a written consent form.
2. 20-60 years old, with clear consciousness, can communicate with the Mandarin and Taiwanese, and are willing to conduct this research.
3. Body mass index according to the Asia Pacific implementation of Bariatric surgery indications, BMI≧37 Kg/m2 or BMI≧32 Kg/m2 combined with metabolic diseases caused by obesity, such as cardiovascular disease, type 2 diabetes, Obstructive Sleep Apnea(OSA), nonalcoholic fatty liver, and degenerative arthritis.
4. Patients with morbid obesity undergoing laparoscopic gastric sleeve resection or laparoscopic gastric bypass surgery.
5. Explain how the smart phone application (Google Fit) and (68 Heart Rate Monitor) are used, and the patient or family member can be operated after returning home.

Exclusion Criteria:

1. After the attending physician evaluates,medical order presentation a person who cannot perform exercise prescriptions.
2. Lower limb limb disorders or amputations cannot coordinate with exercise prescription.
3. Poorly controlled cardiovascular diseases such as arrhythmia, angina, heart failure,myocardial infarction, and chest pain during activities or rest in the past three months.
4. Patients with poor diabetes control, glycosylated hemoglobin (HbA1C) > 9%, with eye lesions or neuropathy.
5. Those with poor blood pressure control, systolic blood pressure greater than 160mmHg or diastolic blood pressure greater than 100mmHg when quiet.
6. Heart rate is greater than 100bpm when quiet.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 85 (Actual)
Dates: Start 2020-01-09 (Actual); Primary Completion 2021-02-23 (Actual); Study Completion 2021-02-23 (Actual)

PRIMARY OUTCOMES:
BMI | baseline(one weeks after recruited)
  using bioelectric impedance(BIA) to measure BMI.the weight in kilograms divided by the square of the height in meters(Kg/m2)
BMI | 1st month after recruited
  using bioelectric impedance(BIA) to measure BMI.the weight in kilograms divided by the square of the height in meters(Kg/m2)
BMI | 2nd month after recruited
  using bioelectric impedance(BIA) to measure BMI.the weight in kilograms divided by the square of the height in meters(Kg/m2)
BMI | 3rd month after recruited
  using bioelectric impedance(BIA) to measure BMI.the weight in kilograms divided by the square of the height in meters(Kg/m2)
objective body composition index | baseline(one weeks after recruited)
  using bioelectric impedance(BIA) to measure body composition
objective body composition index | 1st month after recruited
  using bioelectric impedance(BIA) to measure body composition
objective body composition index | 2nd month after recruited
  using bioelectric impedance(BIA) to measure body composition
objective body composition index | 3rd month after recruited
  using bioelectric impedance(BIA) to measure body composition
Waistline and Waist to hip ratio | baseline(one weeks after recruited)
  using a tape to measure Waistline and Waist to hip ratio.
Waistline and Waist to hip ratio | 1st month after recruited
  using a tape to measure Waistline and Waist to hip ratio.
Waistline and Waist to hip ratio | 2nd month after recruited
  using a tape to measure Waistline and Waist to hip ratio.
Waistline and Waist to hip ratio | 3rd month after recruited
  using a tape to measure Waistline and Waist to hip ratio.

SECONDARY OUTCOMES:
Short Form 36(SF-36) | baseline(one weeks after recruited)
  The SF-36 provides scores for each of the eight health domains and psychometrically-based physical component summary (PCS) and mental component summary (MCS) scores.the scores ranging from 0 to 100. the higher the score, the better the quality of healthy living.
Short Form 36(SF-36) | 1st month after recruited
  The SF-36 provides scores for each of the eight health domains and psychometrically-based physical component summary (PCS) and mental component summary (MCS) scores.the scores ranging from 0 to 100. the higher the score, the better the quality of healthy living.
Short Form 36(SF-36) | 2nd month after recruited
  The SF-36 provides scores for each of the eight health domains and psychometrically-based physical component summary (PCS) and mental component summary (MCS) scores.the scores ranging from 0 to 100. the higher the score, the better the quality of healthy living.
Short Form 36(SF-36) | 3rd month after recruited
  The SF-36 provides scores for each of the eight health domains and psychometrically-based physical component summary (PCS) and mental component summary (MCS) scores.the scores ranging from 0 to 100. the higher the score, the better the quality of healthy living.

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Mei Chen, PhD, Study Chair — alice@ntunhs.edu.tw
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
individual participant data that underline results in a publication
Supporting Information: Study Protocol
Time Frame: starting 12 months after publication
Access Criteria: individual participant data that underline the results reported in this article,after deidentification(test,table,figures,and appendices)

REFERENCES:
- [Result] Robert M, Ferrand-Gaillard C, Disse E, Espalieu P, Simon C, Laville M, Gouillat C, Thivolet C. Predictive factors of type 2 diabetes remission 1 year after bariatric surgery: impact of surgical techniques. Obes Surg. 2013 Jun;23(6):770-5. doi: 10.1007/s11695-013-0868-4. PMID 23355293
- [Result] Janik MR, Rogula T, Bielecka I, Kwiatkowski A, Pasnik K. Quality of Life and Bariatric Surgery: Cross-Sectional Study and Analysis of Factors Influencing Outcome. Obes Surg. 2016 Dec;26(12):2849-2855. doi: 10.1007/s11695-016-2220-2. PMID 27179520
- [Result] Magro DO, Geloneze B, Delfini R, Pareja BC, Callejas F, Pareja JC. Long-term weight regain after gastric bypass: a 5-year prospective study. Obes Surg. 2008 Jun;18(6):648-51. doi: 10.1007/s11695-007-9265-1. Epub 2008 Apr 8. PMID 18392907
- [Result] Woodlief TL, Carnero EA, Standley RA, Distefano G, Anthony SJ, Dubis GS, Jakicic JM, Houmard JA, Coen PM, Goodpaster BH. Dose response of exercise training following roux-en-Y gastric bypass surgery: A randomized trial. Obesity (Silver Spring). 2015 Dec;23(12):2454-61. doi: 10.1002/oby.21332. Epub 2015 Nov 5. PMID 26537198
- [Result] Carnero EA, Dubis GS, Hames KC, Jakicic JM, Houmard JA, Coen PM, Goodpaster BH. Randomized trial reveals that physical activity and energy expenditure are associated with weight and body composition after RYGB. Obesity (Silver Spring). 2017 Jul;25(7):1206-1216. doi: 10.1002/oby.21864. Epub 2017 May 30. PMID 28558160
- [Result] Castello V, Simoes RP, Bassi D, Catai AM, Arena R, Borghi-Silva A. Impact of aerobic exercise training on heart rate variability and functional capacity in obese women after gastric bypass surgery. Obes Surg. 2011 Nov;21(11):1739-49. doi: 10.1007/s11695-010-0319-4. PMID 21104041
- [Result] Campanha-Versiani L, Pereira DAG, Ribeiro-Samora GA, Ramos AV, de Sander Diniz MFH, De Marco LA, Soares MMS. The Effect of a Muscle Weight-Bearing and Aerobic Exercise Program on the Body Composition, Muscular Strength, Biochemical Markers, and Bone Mass of Obese Patients Who Have Undergone Gastric Bypass Surgery. Obes Surg. 2017 Aug;27(8):2129-2137. doi: 10.1007/s11695-017-2618-5. PMID 28285470
- [Result] Kolotkin RL, LaMonte MJ, Litwin S, Crosby RD, Gress RE, Yanowitz FG, Hunt SC, Adams TD. Cardiorespiratory fitness and health-related quality of life in bariatric surgery patients. Obes Surg. 2011 Apr;21(4):457-64. doi: 10.1007/s11695-010-0261-5. PMID 20820940
- See also: Obesity and overweight — http://www.who.int/en/news-room/fact-sheets/detail/obesity-and-Overweight
- See also: Adult obesity empirical guidelines — http://www.hpa.gov.tw/Pages/Detail.aspx?nodeid=1789&pid=10042